CLINICAL TRIAL: NCT03572556
Title: Prospective Descriptive Study of the Angiogenic T Cell Population in Subjects With Hereditary Hemorrhagic Telangiectasia (HHT)
Acronym: TangRO
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: GUILHEM AMRO/AOI 2017
Record Dates: First submitted 2018-06-08; First posted 2018-06-28 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2019-11

CONDITIONS: Hereditary Hemorrhagic Telangiectasia
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Hereditary hemorrhagic telangiectasia patients
  Interventions: Biological: Blood samples; Other: Epistaxis charts
- Controls: Matched for age (+/- 5 ans) and sex.
  Interventions: Biological: Blood samples

INTERVENTIONS:
Biological: Blood samples — * 5 mL dry tube to separate serum
  * Two 6 mL EDTA tubes for plasma separation
  * Eight 6 mL heparinized tubes for flow cytometry (quantification of TANG such as CD3+CD31+CXCR4+ and CEC) and quantification of angiogenesis markers.
Other: Epistaxis charts — Three monthly epistaxis charts to be completed
  Groups: Patients

SUMMARY:
Hereditary hemorrhagic telangiectasia (HHT) results from genetic deregulation of angiogenesis. It is characterized by mucocutaneous telangiectasia responsible for recurrent epistaxis affecting quality of life (anaemia, iron deficiency, social distress). More rarely, HHT is complicated by the appearance of pulmonary, hepatic or cerebral arteriovenous malformations that can lead to serious complications: cerebrovascular accidents, cerebral abscesses, high output heart failure, and massive hemoptysis (1). The intensity of symptoms increases with age but with significant individual variability, even for the same mutation in the same family. Thus, while the mutations responsible for the disease have been identified, the pathophysiology is not fully understood because these mutations do not explain the great diversity of clinical presentations. Other factors not yet identified probably play an important role. Angiogenic T cells (TANG) are a newly individualized T cell population, defined by a CD4+CXCR4+CD31+ phenotype, which plays a key role in differentiating endothelial progenitors (2).

In an earlier study, the investigators showed that patients with HHT had a decrease in CD4+ and CD8+ LT compared to a cohort of healthy subjects (3).

They hypothesize that the lymphopenia mainly involves TANG, whose quantification could make it possible to assess the individual level of angiogenesis during HHT. The evaluation of the TANG levels could thus make it possible to personalize HHT management.

ELIGIBILITY:
Inclusion Criteria:

* Person who has given consent
* Adult
* Person capable of understanding spoken and written French

"Patient" group:

* Certain HHT (3 or 4 Curacao criteria - Appendix 2):
* Recurring epistaxis
* Telangiectasia of the skin or mouth
* Family hereditary context
* Arteriovenous visceral malformations
* Causal mutation identified
* Person capable of completing monthly epistaxis charts

"Control" group :

- Control subjects will be matched to patients for age (+/- 6 years) and sex.

Exclusion Criteria:

* Person not affiliated to a national health insurance scheme
* Pregnant or breastfeeding woman
* Protected adult
* Hemoglobin levels less than 9 g/dl in the last 15 days
* Progressive or recent infectious disease, autoimmune disease or cancer (less than 6 months)
* Immunosuppressive treatment in progress or recent (less than 6 months), including systemic steroid therapy. The use of inhaled or topical steroids is not an exclusion criterion.
* Treatment in progress or stopped less than 6 months ago or to be introduced within the next 3 months of the following medications:

  * bevacizumab
  * tranexamic acid
  * dipeptidyl peptidase 4 inhibitors (diabetic patient)
  * beta-blockers (hypertensive patient)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: outpatient
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2020-05-03 (Actual)

PRIMARY OUTCOMES:
Average monthly duration (in minutes) of epistaxis over the 3 months following inclusion | Through study completion, an average of 3 months
Number/mm3 of circulating TANG (CD3+CXCR4+CD31+) at inclusion. | At inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France